CLINICAL TRIAL: NCT02594982
Title: DANish DELIrium Study On Neurointensive Care Patients. A Two Phase Intervention Study
Brief Title: DANish DELIrium Study On Neurointensive Care Patients
Acronym: DANDELION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsten Moller (Other)
Responsible Party: Sponsor-Investigator, Kirsten Moller, Professor, dept. of Neuroanaesthesiology, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-15007689
Record Dates: First submitted 2015-10-19; First posted 2015-11-03 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2016-10

CONDITIONS: Acquired Brain Injuries; Delirium; Acute Brain Injury
Keywords: Delirium; intensive care nursing; Acute acquired brain injury; neurointensive care; Intensive care delirium screening checklist; Confusion Assessment Method for the ICU
MeSH Terms: conditions — Delirium; Brain Injuries | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention bundle (Other): An intervention bundle consisting of optimized sedation, pain assessment and treatment, early mobilization and sleep.
  Interventions: Other: intervention bundle (sedation, pain, mobilization and sleep)

INTERVENTIONS:
Other: intervention bundle (sedation, pain, mobilization and sleep) — Sedation: Sedation after target RASS Pain: Implementing a pain guideline and CPOT for pain assessment. Mobilization: Implementing a guideline on early mobilization and a daily prescribed mobilization level.
  Sleep: Implementing a daily quite time and changing procedures to minimize noise during the night

SUMMARY:
Abstract Background Studies have shown that delirium in medical and surgical intensive care units (ICUs) increases mortality, length of stay (LOS) as well as the risk of dementia symptoms and cerebral atrophy after discharge. Only few studies have investigated delirium in the neurointensive care unit (N-ICU). Delirium is most often assessed by one of two instruments: Intensive Care Delirium Screening Checklist (ICDSC) or the Confusion Assessment Method for the ICU (CAM-ICU).

Aims

1. To measure the effect of a systematic intervention (sedation, sleep, mobilization and pain) on delirium symptoms in patients with acute acquired brain injury in N-ICU.
2. To validate the ICDSC and CAM-ICU to patients with acute acquired brain injury Method The design of the study is a two-phase interventional trial. Based on a power calculation, 56 patients will be enrolled both in the baseline and the intervention group (n=112).

Part 1: A baseline investigation will be conducted to establish prevalence, duration and type of delirium symptoms in patients with acute acquired brain injury before implementing the intervention bundle.

Part 2: A systematic Intervention protocol will be implemented in the N-ICU. The Intervention elements consist of a sedation, sleep, mobilization and pain treatment regimen based on the newest available evidence.

Enrolled patients will be contacted 12 months after discharge for a follow-up including a quality of life with (EuroQoL-5D) questionnaire, a cognitive test measuring their cognitive end point (Repeatable Battery for Assessment of the Neuropsychological Status) and a short test for dementia symptoms (MMSE, Mini Mental State Examination).

DETAILED DESCRIPTION:
Background It has been established that in medical and surgical intensive care units (ICUs) that delirium increases mortality and length of stay (LOS), as well as the risk of dementia and cerebral atrophy after discharge. There is a lack of studies into delirium in the neurointensive care unit (N-ICU) population, and no studies have addressed the association between delirium, quality of life, dementia symptoms and cerebral atrophy in patients with acquired brain injury after discharge from N-ICU. A recent study has demonstrated a correlation between delirium symptoms in stroke patients and quality of life, and functional levels at 3, 6 and 12 months after N-ICU discharge, suggesting that delirium during the acute phase effects the long-term outcome.

Delirium screening has not been introduced systematically in N-ICUs in Denmark or internationally, and validated instruments are lacking in this population. The Confusion Assessment Method for ICU (CAM-ICU) and the Intensive Care Delirium Screening Checklist (ICDSC) are internationally most recommended and best validated delirium screening tools for non-psychiatric health care staff. Neither of the two instruments, however, has been fully validated in patients with acquired brain injury.

Several studies and guidelines suggest that delirium is potentially preventable by minimizing sedation, and ensuring systematic pain management, early mobilization and adequate sleep. The present study therefore aims to investigate if delirium is preventable in an N-ICU setting by introducing a multi-modal intervention bundle optimizing management of sedation, pain, mobilization and sleep.

Aim

The primary aim of the study:

To measure the effect of the intervention bundle on prevalence, duration and type of delirium symptoms using the Intensive Care Delirium Screening Checklist (ICDSC) and Confusion Assessment Method for the ICU (CAM-ICU) in N-ICU patients with acute acquired brain injury

Secondary aim: To validate ICDSC and CAM-ICU for adult N-ICU with acute acquired brain injury, and investigate if delirium symptoms are negatively correlated with quality of life, cognitive function and dementia symptoms at 12-month follow-up post N-ICU discharge.

Method Study design: A controlled two-phased before-and-after trial. Phase I: Baseline study (4 months), Phase II: Intervention study (4 months). This design was chosen as the most appropriate, because a randomized clinical trial would have a large spill-over effect.

The primary outcome is duration of delirium symptoms with ICDSC and CAM-ICU in the N-ICU based on a hypothesis that it is possible to decrease time with delirium in the N-ICU 20% or more. Power calculation: 56 patients will be enrolled during a 4-month period, in the baseline and the intervention group respectively, yielding a total of 112 patients (20% drop-out rate, 5% significance, 80% power).

Inclusion criteria All Danish speaking adults (18 years or above) with an expected N-ICU length of stay (LOS) more than 48 hours and admitted with acute brain injury from spontaneous or traumatic bleeding, such as subarachnoid hemorrhage (SAH), intracranial hemorrhage (ICH) or traumatic brain injury (TBI).

Exclusion criteria Patients not expected to survive 48 hours, or continues Richmond Agitation-Sedation Score (RASS) of -4 or -5 during the stay in the N-ICU.

Data collection Demographics: age, gender, primary diagnosis, marital status and living situation, education, BMI, and alcohol consumption. Clinical data include: Glasgow Coma Score (GCS), Richmond Agitation and Sedation Scale (RASS), ICDSC, CAM-ICU, Acute Physiology and Chronic Health Evaluation II (APACHE II), Simplified Acute Physiology Score (SAPS II), intubation status, sedation agent and dose, type of mobilization and pain status. Follow-up includes EuroQoL-5D (EQ-5D), Repeatable Battery for Assessment for the Neuropsychological Status (RBANS) and Mini Mental State Examination (MMSE) questionnaire at 12 months after discharge.

Phase I Baseline study (4 months). A baseline investigation will be conducted to establish the prevalence, duration and type of delirium symptoms in patients with acute acquired brain injury. Usual care will be provided at this time. For validation a psychiatric team will rate included patients usingThe Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) and The International Classification of Diseases (ICD-10) as the gold standard. The psychiatric team assesses patients the first and second day after the patient has a RASS -2 or above for 24 hours.

Phase II Intervention study (4 months). After full implementation of the intervention bundle, the study will be conducted to establish the prevalence, duration and type of delirium symptoms in patients with acute acquired brain injury. The psychiatric team assesses patients the first and second day after the patient has a RASS -2 or above for 24 hours.

Implementation of intervention An all day workshop introducing the multi-modal intervention bundle will be held for all nurses in the unit. The study nurses will be specially trained to maintain study protocol. Physicians will be informed and trained on a weekly morning meeting during phase II, and some will participate in the all day workshop. Journal audits will be used as monitoring the implementation. The Intervention bundle consist of a sedation, sleep, mobilization and pain treatment regimen based on the newest available evidence in the four areas.

Sedation: Sedatives will be kept to a minimum by daily orders for target RASS sedation level and titration of sedatives by primary nurse. Dose and agent will be recorded.

Sleep: Sleep will be optimized by systematic use of earplugs at night, dim lighting, visitation restrictions, and midday rest periods. Procedures (e.g. blood samples) will be carried out in the day time instead of night time. Hours of activity/rest will be assessed by an actiwatch (actigraph).

Pain: A strategy of multi-modal pain management combining pharmacological and non-pharmacological interventions will be implemented. Pain will be assessed by Critical-Care Pain Observation Tool (CPOT) for unresponsive patients and Numeric Rating Scale (NRS) for patient-reported pain.

Mobilization: Systematic early mobilization will be implemented by daily orders for mobilization level and a mobilization guideline.

Follow-up: Follow-up will be conducted on all possible patients in the two study groups at twelve months post N-ICU discharge. Patients will come to the hospital for the EQ-5D for self-rated health, RBANS for cognitive function and the MMSE questionnaire for dementia symptoms.

Ethical considerations The study includes an observational and an interventional part introducing optimized treatment and care according to current best international evidence. The intervention items will be implemented in the entire unit as standard care for all patients. Most patients will be unable to give initial consent to the study due to their cerebral status. Relatives and general practitioner will be contacted and informed verbally and in writing to provide consent by proxy. The study is approved by the Regional and national ethics committees and the Danish Data Protection Agency.

Data analysis Prevalence, type and duration of delirium symptoms in the baseline group will be compared to the intervention group. Furthermore the two groups will be compared on LOS and mortality. Patients ICDSC score are compared with EQ-5D, RBANS and MMSE in order to investigate possible associations between delirium and self-rated health, cognitive function and dementia.

All data will be coded and plotted in Excel and SPSS for the statistical data analysis. Hardware and worksheets are handled and stored as prescribed by the Danish Data Protection Agency. There will be used descriptive and analytical statistics. Categorical variables will be described as frequency and percent. Continuous variables will be described as mean and standard deviation (SD). The two groups will be compared by correlation analysis, univariate and multivariate regression analyzes and questionnaires are analyzed by a paired t-test to compare the two groups' average score.

ELIGIBILITY:
Inclusion Criteria:

* All Danish speaking adults (18 years or above)
* Expected N-ICU length of stay (LOS) more than 48 hours
* Admitted with acute brain injury from subarachnoid hemorrhage (SAH), intracranial hemorrhage (ICH) or traumatic brain injury (TBI).

Exclusion Criteria:

* Patients not expected to survive 48 hours
* Richmond Agitation-Sedation Score (RASS) of -4 or -5 during the stay in the N-ICU.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Duration of delirium symptoms. | Minimum 48 hours and up to 4 weeks
  Patients are assessed two times per day for delirium symptoms with ICDSC and the CAM-ICU during their stay on the N-ICU. duration of delirium symptoms measured by CAM-ICU and ICDSC will be analysed individually and the one with the best performance test will be presented as the primary outcome measure.

SECONDARY OUTCOMES:
Validation of ICDSC and CAM-ICU | 2 days. On the first and second assessable day (RASS -2 or above).
  Investigate sensitivity and specificity of ICDSC and CAM-ICU. A psychiatric team assess patients with diagnostic criteria DSM-V and ICD-10. Laura Krone Larsen and nurses assess patient with the ICDSC and the CAM-ICU for comparison with the psychiatric assessment.
Prevalence of delirium symptoms | 1 day and up to 4 weeks.
  During baseline (phase 1) and the intervention phase (phase 2) patients are assessed twice daily for delirium symptoms with the ICDSC and CAM-ICU.
Length of Stay | 2 days (48 hours) and up til 4 weeks
  LOS is compared between the baseline (phase 1) and the intervention phase (phase 2)
Quality of life after 12 month after discharge | 12 month
  12 month after discharge patients are assess with EQ-5D.
Mortality | 1 year
  Mortality up til one year after discharge is compared between the baseline (phase 1) and the intervention phase (phase 2)
cognitive function after 12 month after discharge | 12 month
  12 month after discharge patients are assess with RBANS.
Type of delirium symptoms | 1 day (24 hours) and up to 4 weeks.
  Hyper, hypo or mixed delirium symptoms assessed with RASS and in words by Laura Krone Larsen and Nurses. Comments and descriptions on delirium symptoms are collected during phase 1 and phase 2.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten moeller, professor, Principal Investigator — Rigshospitalet, 2093
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Sealand, Denmark

REFERENCES:
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Gelinas C, Fillion L, Puntillo KA, Viens C, Fortier M. Validation of the critical-care pain observation tool in adult patients. Am J Crit Care. 2006 Jul;15(4):420-7. PMID 16823021
- [Background] Kamdar BB, King LM, Collop NA, Sakamuri S, Colantuoni E, Neufeld KJ, Bienvenu OJ, Rowden AM, Touradji P, Brower RG, Needham DM. The effect of a quality improvement intervention on perceived sleep quality and cognition in a medical ICU. Crit Care Med. 2013 Mar;41(3):800-9. doi: 10.1097/CCM.0b013e3182746442. PMID 23314584
- [Background] Morandi A, Brummel NE, Ely EW. Sedation, delirium and mechanical ventilation: the 'ABCDE' approach. Curr Opin Crit Care. 2011 Feb;17(1):43-9. doi: 10.1097/MCC.0b013e3283427243. PMID 21169829
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Naidech AM, Beaumont JL, Rosenberg NF, Maas MB, Kosteva AR, Ault ML, Cella D, Ely EW. Intracerebral hemorrhage and delirium symptoms. Length of stay, function, and quality of life in a 114-patient cohort. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1331-7. doi: 10.1164/rccm.201307-1256OC. PMID 24102675
- [Background] Olson DM, Borel CO, Laskowitz DT, Moore DT, McConnell ES. Quiet time: a nursing intervention to promote sleep in neurocritical care units. Am J Crit Care. 2001 Mar;10(2):74-8. PMID 11244674
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Svenningsen H, Tonnesen E. Delirium incidents in three Danish intensive care units. Nurs Crit Care. 2011 Jul-Aug;16(4):186-92. doi: 10.1111/j.1478-5153.2011.00421.x. PMID 21651659
- [Background] Yu A, Teitelbaum J, Scott J, Gesin G, Russell B, Huynh T, Skrobik Y. Evaluating pain, sedation, and delirium in the neurologically critically ill-feasibility and reliability of standardized tools: a multi-institutional study. Crit Care Med. 2013 Aug;41(8):2002-7. doi: 10.1097/CCM.0b013e31828e96c0. PMID 23863231
- [Derived] Larsen LK, Frokjaer VG, Nielsen JS, Skrobik Y, Winkler Y, Moller K, Petersen M, Egerod I. Delirium assessment in neuro-critically ill patients: A validation study. Acta Anaesthesiol Scand. 2019 Mar;63(3):352-359. doi: 10.1111/aas.13270. Epub 2018 Oct 16. PMID 30324653